CLINICAL TRIAL: NCT03367689
Title: A Two-stage Simon Design Phase II Study for NOn-BRCA Metastatic BReast Cancer (MBC) Patients With Homologous Recombination Deficiency Treated With OLAparib Single Agent
Brief Title: A Two-stage Simon Design Phase II Study for Non-BRCA MBC Patients With HRD Treated With Olaparib Single Agent
Acronym: NOBROLA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very slow recruitment due to subject profile
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP100; 2016-002892-80 (EudraCT Number)
Record Dates: First submitted 2017-11-24; First posted 2017-12-11 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: This is an international, multi-centre, non-controlled, open-label, single arm, two-stage Simon Design phase II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib 300 mg (Experimental): Patients whose tumours are identified as Homologous Recombination Deficient, will receive olaparib 300 mg (two tablets of 150mg) orally twice daily (bid) on days 1-28 each 28 days.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib 300 mg twice a day (orally) beginning on Day 1 and continuing through Day 28 of every 28-day cycle.
  Other Names: Lynparza; AZD2281

SUMMARY:
This is an international, multi-centre, non-controlled, open-label, single arm, two-stage Simon Design phase II study for non-BRCA metastatic breast cancer (MBC) patients with homologous recombination deficiency treated with Olaparib single agent.

The main objective is to assess the efficacy of olaparib single agent as determined by Clinical Benefit Rate (CBR) using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

In the first stage Triple negative (TN) non-BRCA, metastatic breast cancer (MBC) patients whose tumours exhibited any characteristic related to homologous recombination deficiency (HRD). In the second stage, luminal patients (RH positive HER2 negative) will be allowed in the same conditions that TN.

Patients whose tumours are identified as Homologous Recombination Deficient by deleterious HRR gene mutations (according to Foundation Medicine's Foundation One assay) will receive olaparib 300 mg (two tablets of 150mg) orally twice daily (bid) on days 1-28 each 28 days.

Study commitment is 39 patients: 17 patients will be enrolled at first stage and 22 at the second stage.

The total duration of the study period is 34 months.

DETAILED DESCRIPTION:
This is an international, multi-centre, non-controlled, open-label, single arm, two-stage Simon Design phase II study for non-BRCA metastatic breast cancer (MBC) patients with homologous recombination deficiency treated with Olaparib single agent.

The main objective is to assess the efficacy of olaparib single agent as determined by Clinical Benefit Rate (CBR) using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

Triple negative non-BRCA metastatic breast cancer women (for the first stage) age ≥ 18 years that had previously received at least one (and no more than three) line for their metastatic disease. Patients must have previously received taxanes either in the early or in the metastatic scenario. To be included in the trial, tumours must be considered homologous recombination deficient (HRD) according to Foundation Medicine's Foundation One assay. Evidence of measurable metastatic disease is required.

In the second stage, luminal patients (RH positive HER2 negative) will be allowed to participate in the same conditions that TN patients.

Patients whose tumours are identified as Homologous Recombination Deficient by deleterious HRR gene mutations (according to Foundation Medicine's Foundation One assay) will receive olaparib 300 mg (two tablets of 150mg) orally twice daily (bid) on days 1-28 each 28 days.

Study commitment is 39 patients: 17 patients will be enrolled at first stage and 22 at the second stage.

During the period between the end of the first stage and the beginning of the second, an interim analysis will be conducted to assess the viability of the second part of the trial.

The total duration of the study period is 34 months.

Stage I:

* Recruitment period: 10 months
* Follow-up period: Up to 6 months after last patient included in the study

Stage II:

* Recruitment period: 12 months
* Follow-up period: up to 6 months after last patient included in the study

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for inclusion only if they meet ALL the following criteria:

1. Female patients ≥ 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) score lower or equal to 1.
3. Life expectancy greater or equal to 16 weeks.
4. Confirmed TN locally advanced or metastatic breast cancer in the first stage. For the second stage, luminal-like patients (RH-positive HER2-negative) will be allowed.
5. Wild type BRCA1 and BRCA2 (germline). Variants with unknown significance are eligible.
6. Tumors must exhibit a HRD signature according to Foundation Medicine's Foundation One assay. Formalin fixed, paraffin embedded (FFPE) tumor sample from the metastatic cancer must be available for central testing. If there is not written confirmation of the availability of an archived tumor sample prior to enrolment the patient is not eligible for the study.
7. No more than three (and at least one) previous lines for the metastatic disease. Previous treatment must include taxanes (neo/adjuvant scenario is also possible) if not formally contraindicated.
8. Patient must have measurable disease according to RECIST 1.1 criteria. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis > or equal 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
9. Patients must have normal organ and bone marrow function measured within 35 days prior to administration of study treatment as defined below:

   Hematological: White blood cell (WBC) count >3.0 x 109/L, absolute neutrophil count (ANC) > or equal 1.5 x 109/L, platelet count ≥100.0 x109/L, and hemoglobin >10.0 g/dL (>6.2 mmol/L) with no blood transfusion in the past 35 days.

   Hepatic: bilirubin ≤ 1.5 times the upper limit of normal (x ULN); alkaline phosphatase (ALP), Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) < or equal 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be < or equal 5x ULN.

   Renal: creatinine clearance estimated using the Cockcroft-Gault equation of > or equal 51 mL/min
10. Patient has been informed about the nature of study, and has agreed to participate, and signed the Informed Consent form (ICF) prior to participation in any study-related activities
11. No other malignancies within the past five years except adequate treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
12. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCICTCAE version 4.03 Grade < or equal 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
13. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days prior to administration of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as:

Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments; Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50; Radiation-induced oophorectomy with last menses >1 year ago; Chemotherapy-induced menopause with >1 year interval since last menses; Surgical sterilization (bilateral oophorectomy or hysterectomy).

Exclusion Criteria:

Patients will be excluded from the study if they meet ANY of the following criteria:

1. RH-positive (based on local laboratory results) or unknown for the first stage. In the second stage, luminal-like HER2-negative patients will be allowed.
2. HER2-positive (based on local laboratory results [performed by immunohistochemistry/fluorescence in situ hybridization (FISH)] or unknown.
3. Locally advanced breast cancer candidate for a radical treatment.
4. Has deleterious germline BRCA1 or BRCA2 mutation as determined by local test.
5. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 35 days.
6. Patients with symptomatic visceral disease are not eligible.
7. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years.
8. Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML
9. Have had a major surgery (defined as requiring general anesthesia) or significant traumatic injury within 2 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery or patients that may require major surgery during the course of the study.
10. Resting ECG with QTc > 470 msec on 2 or more time points within a 24-hour period or family history of long QT syndrome.
11. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
12. Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors. The required washout period prior to starting olaparib is 2 weeks.
13. Concomitant use of known strong or moderate CYP3A inducers. The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
14. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
15. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
16. Patients with known active hepatitis (i.e. Hepatitis B or C).
17. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
18. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.9).
19. Are unable to swallow orally administered medication.
20. Patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
21. Chronic daily treatment with corticosteroids with a dose of ≥ 10mg/day methylprednisolone equivalent (excluding inhaled steroids), except for prophylaxis use.
22. Female patients who are pregnant or breastfeeding, or adults of reproductive potential who are not using effective birth control methods.
23. Patients unwilling to or unable to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
24. Patients that have previously receive any PARP inhibitor for any reason, including olaparib.
25. Known hypersensitivity to olaparib excipients or any of the excipients of the product.
26. Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site).
27. Previous enrolment in the present study.
28. Participation in another clinical study with an investigational product during the last 3 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of olaparib single agent in non-BRCA MBC patients whose tumours exhibit an homologous recombination deficiency (HRD) signature, as determined by Clinical Benefit Rate (CBR) using RECIST 1.1 criteria | Baseline up to 24 weeks
  The CBR as best response, defined as the percentage of patients who experience a complete response, partial response or stable disease for at least 24 weeks and assessed by modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) criteria

SECONDARY OUTCOMES:
To assess the accuracy of Foundation One's HRR assay in predicting the proportion of patients with response to olaparib. | Baseline up to 34 months
  The positive predictive value (PPV) of the signature to predict patients that achieved objective response and clinical benefit.
To assess incidence of Treatment-Emergent Adverse Events (Safety profile) of olaparib in this population | Baseline up to 34 months
  This study will consider the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v4.03 criteria) grade 3 and 4 events (AEs) and serious AEs (SAEs) in order to assess the safety and tolerability objectives.
To investigate the prevalence of HRD signature within triple negative and luminal non-BRCA patients' cohorts | Baseline up to 34 months
  The percentage of patients with HRD according to the Foundation Medicine's Foundation One assay within triple negative and luminal (in the second stage) non-BRCA patients' cohorts
To explore the efficacy of olaparib in terms of Progression-free survival (PFS) | Baseline up to 34 months
  The PFS defined as the time from the first dose of study drugs until objective tumour progression or death, as assessed by the investigator per RECIST v1.1.
To explore the efficacy of olaparib in terms of objective response rate (ORR) | Baseline up to 34 months
  The ORR defined as the proportion of patients with best objective response of confirmed complete response (CR) or partial response (PR) according to RECIST criteria guidelines (version 1.1).
To explore the efficacy of olaparib in terms of overall survival (OS) | Baseline up to 34 months
  The OS defined as the time from the first dose of study drugs until death from any cause or the last date the patient was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortes, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (5):
- Spain (5):
  - Hospital del Mar, Barcelona
  - Onkologikoa, Donostia / San Sebastian
  - Institut Català d' Oncologia L'Hospitalet (ICO), L'Hospitalet de Llobregat
  - Hospital Ramón y Cajal, Madrid
  - Hospital Arnau de Vilanova de Valencia, Valencia

REFERENCES:
- [Derived] Cortes A, Lopez-Miranda E, Fernandez-Ortega A, Caranana V, Servitja S, Urruticoechea A, Lema-Roso L, Marquez A, Lazaris A, Alcala-Lopez D, Mina L, Gener P, Rodriguez-Morato J, Antonarelli G, Llombart-Cussac A, Perez-Garcia J, Cortes J. Olaparib monotherapy in advanced triple-negative breast cancer patients with homologous recombination deficiency and without germline mutations in BRCA1/2: The NOBROLA phase 2 study. Breast. 2024 Dec;78:103834. doi: 10.1016/j.breast.2024.103834. Epub 2024 Nov 3. PMID 39520738